CLINICAL TRIAL: NCT00433056
Title: Strategic, Long Term, Immunologically Driven Treatment Interruptions in Patients on Effective HAART: A Controlled, Randomized Study
Brief Title: Long Term Treatment Interruptions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOTTI
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infections; AIDS
Keywords: STI; HIV; CD4; HIV-RNA; HAART
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

ARMS (2):
- 1 (Experimental): STI
  Interventions: Other: STI
- 2 (Active Comparator): stable HAART, Any registered regimen containing NRTIs (AZT or D4T or 3TC or TDF or DDI), NNRTIs (EFV or NVP) or PIs (RTV-boosted ATV; IDV; LPV, fosAPV, SQV; unboosted ATV or NFV)is allowed according to international guidelines
  Interventions: Drug: stable HAART

INTERVENTIONS:
Other: STI — CD4 guided treatment interruption
  Arms: 1
Drug: stable HAART — continuous therapy
  Arms: 2

SUMMARY:
LOTTI study Centers

This a multicenter, multinational study.

Clinical phase: III

Objectives

The primary objective is to compare efficacy and safety of continuing a conventional HAART in chronically infected HIV patients with a therapeutic strategy based on long term, immunologically driven treatment interruptions.

Secondary objectives are:

* To verify the risk of developing viral resistance
* To verify the effect of the two strategies on metabolic parameters
* To verify the possibility to steadily discontinue antiretroviral therapy in patients who started it with baseline immunological values higher than those currently recommended by international guidelines for HIV treatment
* To identify predictive variables of the possibility to safely discontinue antiretroviral therapy
* To verify the dynamic of CD4+ cell loss and HIV replication after treatment interruption

Number of Patients: A total of 320 patients.

Study design:

Controlled, Randomized, Open study The study will last 5 years

Treatment arms:

Patients will be randomized in a ratio 1:1 to one of the two treatment arms Control group continuing the ongoing therapy STI group performing long term CD4 guided structured treatment interruptions In the STI arm patients will stay off therapy until their CD4 count will drop < 350 cells/mcL (one measurement will be considered sufficient). At that time point patients will resume the HAART regimen they were assuming before STI and will continue HAART until they CD4 count will raise > 600 cells/mcL (at least 2 consecutive measurements 2 months apart) and their HIV-RNA will drop below the detection limit of 50 copies/ml (one measurement will be considered sufficient). When both the CD4 count and the viral load will be within these pre-set values they will stop therapy again. There is no limit to the number of interruptions and re-start cycles during the study period

End points:

The primary end-point for the evaluation of the main objective of the study will be clinical. The primary outcome measure will be based on the occurrence of a clinical end-point defined as: disease progression (occurrence of any AIDS defining event), death for any cause or the occurrence of clinical events requiring hospital admission

The secondary objectives of the study will be evaluated on the basis of:

* Mean variation of blood cholesterol and triglycerides from baseline values.
* Development of lipodystrophy or modification of a pre-existing lipodystrophy
* Time off therapy.
* Variation of CD4 counts and HIV-RNA levels
* Genotypic tests to be performed in the case of HIV-RNA > 1000 copies/ml while on therapy for at least 4 months or one month after each treatment interruption.

Statistics:

The study is powered to evaluate equivalence between the two strategies under the assumption that, in the control arm, the primary end-point would be observed in a proportion of subjects < 7% and that the same proportion in the STI arm would not exceed 10% with a maximum allowed 95%CI of 12%. 320 patients will be needed for alfa = 5% and 1-beta = 80%. The primary analysis will be made according to the intention-to-treat approach and therefore no correction for eventual drop outs is needed. In addition, a secondary per-protocol analysis will be performed.

DETAILED DESCRIPTION:
Rationale

As the current regimens cannot eradicate HIV infection, persons living with HIV are doomed to assume chronic therapies with often very demanding daily schedules. In the long run, this may lead to reduced adherence to therapy, to incomplete suppression of viral replication and to the emergence of resistant viruses that can vanish the patients' efforts. Furthermore with continued exposure to antiretroviral drugs, patients have begun to experience new adverse effects including body fat redistribution, dislipidemia, diabetes, insulin resistance, osteopenia and the fear of unexpected complications such as cardiovascular diseases has raised. A variety of strategies has emerged to try to help the long-term management of HAART. Researchers have focused their attention on the development of simpler regimens. An alternative approach involves various types of structured treatment interruptions (STI). Several different roles have been claimed for STIs. They have been postulated to enhance specific immune response and allow control of viral replication, in the absence of continuous HAART, in seroconverters. In advanced treatment failures STIs has been suggested to favor the overgrowth of wild-type virus in the peripheral circulation and thus facilitate the "disappearance" of resistance mutations. In chronically infected patients without virologic failure STIs have been explored to boost HIV specific immune responses and, more recently, to reduce drug exposure, promote adherence and minimize drug-related morbidity .

Various strategies with fixed intervals for on and off periods, or with specific thresholds, either immunologic or virologic, for re-initiation of therapy have been explored.

To date, unanswered questions about STIs or even pulse therapy include the risk of exposing patients to differential drug levels which may enhance selection of resistant mutants, the effects of re-seeding of viral reservoirs, the real extent of the assumption that less drug is associated with less toxicity or better adherence, and the overall outcome compared to continuous HAART.

Finally STIs and pulse therapy may result strictly linked with questions raised by new treatment recommendations: what to do with individuals who began therapy at a CD4 + cell level above the currently recommended threshold, and how to manage those patients who, under HAART, have gained a CD4 cell count far above this threshold.

We will conduct a controlled, prospective and randomized trial on a cohort of chronically HIV infected individuals on effective HAART to address most of these open questions. We will apply an individualized pulse therapy strategy, driven by CD4 + cell count, and will compare it with conventional continuous HAART.

Study objectives

Primary objective of the study is:

To compare efficacy and safety of continuing a conventional HAART in chronically infected HIV patients with a therapeutic strategy based on long term, immunologically driven treatment interruptions.

Secondary objectives are:

* To verify the risk of developing viral resistance
* To verify the effect of the two strategies on metabolic parameters
* To verify the possibility to steadily discontinue antiretroviral therapy in patients that started it with baseline immunological values higher than those currently recommended by international guidelines for HIV treatment
* To identify predictive variables of the possibility to safely discontinue antiretroviral therapy
* To verify the dynamic of CD4 + loss and HIV replication after treatment interruption

As the study wants to enroll patients strictly reflecting the population of HIV infected individuals, previous mono or dual therapies as well as the presence of co-morbidities such as HBV and HCV co-infection do not constitute exclusion criteria, but will be recorded.

Study design

This is a multicenter, randomized, controlled, open, comparative study. The trial will have a follow-up of 5 years.

Patients will be monitored according to the international and local guidelines for HIV infection as far as timing and type of laboratory and clinical controls. Laboratory exams will be decided locally and only a few key tests are required for the study. The timing of laboratory evaluation will be 1 and 2 months after each treatment interruption and thereafter every 2 months in the STI arm and every 4 months in the control group. All data will be stored in a computerized data-base.

Study arms and management of the study

Patients will be randomized in the ratio 1: 2 to one of the following treatment arms:

1. Continuing their ongoing HAART (control)
2. Long term treatment interruption (STI)

Randomization will be accomplished centrally according to a pre-determined, computer-generated random list.

In the control group, patients will be allowed to change therapy for virological, toxicological or personal reasons. All variation will be recorded. Patients changing therapy will be still included in the ITT analysis, but will be considered failures in the AT analysis. Patients stopping therapy, for any reason and not resuming it within 3 months will be considered as failures for both the ITT and AT analysis In the STI arm, patients will stay off therapy until their CD4 count drop < 350 cells/mcL (one measurement will be considered sufficient). At that time point patients will resume the HAART regimen they were assuming before the STI period and will continue HAART until their CD4 count raises > 600 cells/mcL and their plasma HIV-RNA drops below the detection limit of 50 copies/ml (one measurement will be considered sufficient). When both the CD4 count and the viral load will be within these pre-set values they will stop therapy again. There is no limit to the number of interruptions and re-start cycles during the study period 160 patients will be allocated in the STI arm and 80 patients in the control arm.

End points and evaluation criteria

The primary end-point for the evaluation of the main objective of the study will be clinical:

The primary outcome measure will be based on the occurrence of a clinical end-point defined as: disease progression (occurrence of any AIDS defining event), death for any cause or the occurrence of clinical events requiring hospital admission

The secondary objectives of the study will be evaluated on the basis of:

* Mean variation of blood cholesterol and triglycerides from baseline values. Development of lipodystrophy or modification of a pre-existing lipodystrophy
* Time off therapy, variation of CD4 counts and HIV-RNA levels
* Genotypic tests to be performed in the case of HIV-RNA > 1000 copies/ml while on therapy for at least 4 months or one month after each treatment interruption.

Duration of the study

Treatment will be continued for 5 years under the study conditions. Patients completing the study period and still responding to therapy will be kept on the same regimen.

Statistical evaluation of the study will be performed yearly. A first interim analysis will be performed when the mean follow-up will reach 3 years.

Monitoring

Laboratory tests during the study period will be performed in he fasting state. The following tests and procedures are required and will be recorded in the electronic data base. It is also advised to perform on regular basis haemogram, renal function tests, blood glucose and amylase. Other test could be performed according to local needs or particular situations related to the specific management of single patients:

Baseline (all patients)

1) Informed consent and treatment randomization 2) Biochemical analysis: ALT, AST, total cholesterol and HDL, triglycerides 3) CD4 count, CD8 count 4) Plasma HIV-RNA 5) Clinical evaluation, anamnestic and demographic data: sex, age, risk factor for HIV infection, CDC AIDS classification, time on ART, time on current HAART, previous antiretroviral drugs, previous sub-optimal ARTs, current antiretroviral drugs, presence and grade of lipodystrophy, time with HIV-RNA below detection, nadir CD4, CD4 at start of antiretroviral therapy.

1. month after each STI (only STI group) 1) CD4 count, CD8 count
2. months after each STI (only STI group) 1) Biochemical analysis: ALT, AST, cholesterol (total and HDL), triglycerides 2) CD4 count, CD8 count 3) Plasma HIV-RNA, Genotype 4) Clinical evaluation: disease progression, lipodystrophy assessment

Every 2 months thereafter (STI group) or every 4 months from baseline (control group)

1. Biochemical analysis: ALT, AST, cholesterol (total and HDL), triglycerides
2. CD4 count, CD8 count
3. Plasma HIV-RNA
4. Clinical evaluation: disease progression, lipodystrophy assessment

Additional tests

Additional tests will be requested in specific cases:

1. a second genotype after 4 months from the initiation of the STI period will be performed in all patients showing a major mutation in the genotype performed 2 months after STI start
2. a genotype will be performed in all patients either in the STI or in the control group showing a viral load above 1000 copies/ml after a continuous treatment period (on drugs) > 4 months.

Statistical considerations

The study is powered to evaluate equivalence between the two strategies under the assumption that, in the control arm, the primary end-point would be observed in a proportion of subjects < 7% and that the same proportion in the STI arm would not exceed 10% with a maximum allowed 95%CI of 12%. According to the model published in Controlled Clinical Trials 1982; 3: 345-353,320 patients will be needed for alfa = 5% and 1-beta = 80%.

The primary analysis will be made according to the intention-to-treat approach and therefore no correction for eventual drop outs is needed.

In addition, a secondary per-protocol analysis will be performed. Chi-square or Fisher's exact test that will be used to analyze all categorical variables. Time to treatment failure will be estimated using Kaplan-Meier product-limit estimates (that will be presented graphically). The log-rank test will be used to assess the difference between the survival curves for each arm, while ANOVA test and Student's t test will be used for continuous variables unless the variables will not be normally distributed, in which case the Kruskal-Wallis and Mann-Whitney U tests will be used. Logistic regression analysis (forward stepwise model) will be used to evaluate the relationship between variables and outcome.

All tests will be two-sided and a P value inferior to 0.05 will be regarded as significant.

The analysis of data will be performed by the proposing Study Center with the SPSS statistical software package for Windows, version 13.0.

Drugs

This is a spontaneous study. It is proposed that all drugs will be dispensed according to standard procedures.

Data use

Data will be used for scientific porpoises only. The analysis will be performed yearly and the results will be disclosed to the major participating groups for discussion and comments. The type and timing of publication of data will be agreed among the participants to the study. The authorship of each presentation will be agreed among participants. It is foreseeable that no more than 10 authors will be included for each publication. The number of authors for each group will be proportional to the number of patients included at the site. All participants will be acknowledged as members of the study group. The principal investigator at each site will be responsible for indicating the researchers to include as authors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years
* Informed consent signed
* Effective ongoing treatment (HIV-RNA < 50 copies/ml). Treatment must be based on any triple drug therapy. Patients must be on the same steady therapy for at least 3 months.
* Current CD4 cell count above 600 cells/mcL and nadir of CD4 cell count > 200 cells/mcL

Exclusion Criteria:

* Childbearing or breastfeeding. Women of childbearing potential will be asked to adopt effective contraceptive methods or behaviors
* Any ongoing grade 4 (WHO) AE or laboratory abnormality with the exclusion of cholesterol, triglycerides for which a grade 3 (AHA) level will be considered an exclusion criteria.
* Previous diagnosis of AIDS
* Patients with HBV coinfection on active anti-HIV treatment with either lamivudine and/or tenofovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2004-01

PRIMARY OUTCOMES:
The primary outcome will be clinical response: Death, ADE, pathology requiring hospital admission | 5 years

SECONDARY OUTCOMES:
Mean variation of blood cholesterol and triglycerides from baseline values. Development of lipodystrophy or modification of a pre-existing lipodystrophy | 5 years
Time off therapy, variation of CD4 counts and HIV-RNA levels | 5 years
Genotypic tests to be performed in the case of HIV-RNA > 1000 copies/ml while on therapy for at least 4 months or one month after each treatment interruption. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Franco Maggiolo, MD, Principal Investigator — Ospedali Riuniti, Bergamo
Locations (1):
- Ospedali Riuniti, Bergamo, BG, Italy